CLINICAL TRIAL: NCT05038345
Title: Inpatient Care Utilization and Epidemiology of Hirschsprung Disease in the United States: Analysis of the National Inpatient Sample
Brief Title: Hirschsprung Disease Trends in the United States: Analysis of the National Inpatient Sample
Status: Terminated | Type: Observational
Why Stopped: Per PI, the study was terminated prematurely since the data collection was completed
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Rajmohan Dharmaraj, MD Assistant Professor, University of New Mexico
Other Study IDs: 18-697
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pull through surgery — The principal purpose of pull through surgery for Hirschsprung disease is to remove aganglionic bowel and reconstruct the intestinal tract by connecting the normally innervated bowel just above the anus so that normal sphincter function is preserved.

SUMMARY:
Hirschsprung disease (HD) is associated with significant morbidities including long-term bowel dysfunction. The aim of this study was to update national and regional trends in the epidemiology and inpatient care utilization of HD in the United States between 2009 and 2014 using the National Inpatient Sample (NIS).

DETAILED DESCRIPTION:
Hirschsprung disease (HD) is a congenital condition characterized by the absence of ganglion cells in the myenteric and submucosal plexuses of the distal intestine, which results in lack of peristalsis and functional intestinal obstruction. The aganglionosis involves the rectum or rectosigmoid in most cases, but it can extend for varying lengths, and in 5-10% of cases can involve the entire colon or even a significant amount of the small intestine. The incidence of this disease is approximately 1 in 5000 live births and is approximately three times more common in males. HD is a multifactorial disease caused by both genetic and environmental factors, and HD may also be part of a syndrome, most commonly Trisomy 21.

The principal purpose of surgical management of HD is to remove aganglionic bowel and reconstruct the intestinal tract by connecting the normally innervated bowel just above the anus so that normal sphincter function is preserved. Over the last decades, surgical management has changed from original three-stage approach to recent introduction of minimally invasive one-stage procedures, which appears to be safe, and facilitates early feeding and discharge. Although surgical treatment definitively removes the histologically defined pathological intestinal segment, many patients with HD continue to experience bowel dysfunction, obstructive symptoms and recurrent enterocolitis requiring frequent hospitalizations.

Huang et al had shown that HD discharges, associated demographics, and numbers of pull-through procedures remained stable from 1997 to 2006. There is a paucity in the literature regarding cost components associated with care of hospitalized patients with the primary diagnosis of HD. An information update regarding inpatient care utilization for HD is needed to better understand current HD disease burden and inpatient care practice. The primary objective of this study was to analyze cost of HD-related admissions in the United States between 2009 and 2014 using the National Inpatient Sample (NIS) database. Secondary objectives were to update national and regional trends in the epidemiology of HD related hospital utilization, and to examine changing demographics, hospital mortality and length of hospital stay (LOS) in these HD patients.

ELIGIBILITY:
Inclusion Criteria:

* We included all patients who were 18 years or younger with an ICD-9-CM code of 751.3 for HD among the first 10 diagnosis.

Exclusion Criteria:

* Data from 2015 to 2018 were not included since diagnoses and procedures were reported using the ICD-10-CM coding system.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: We included all patients who were 18 years or younger with an ICD-9-CM code of 751.3 for HD among the first 10 diagnosis. Patients whose discharge disposition was transfer to another hospital were excluded to avoid over-counting. We identified patients with a pull-through procedure using following ICD-9-CM codes: 4592, 4593, 4594, 4595, 4840, 4841, 4842, 4843, 4849, and 4865. We tracked the number of these pull-through procedures a patient received. We used all 15 procedure codes to identify pull-through procedures and other procedures. To identify common discharge diagnoses we used the first five diagnosis codes. To identify congenital anomalies we used all diagnosis codes.
Sampling Method: Probability Sample
Enrollment: 2787 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to analyze cost of HD-related admissions in the United States between 2009 and 2014 using the National Inpatient Sample (NIS) database. | 2009 to 2014.

CONTACTS AND LOCATIONS:
Overall Officials: Yiliang Zhu, Study Director — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang EY, Tolley EA, Blakely ML, Langham MR. Changes in hospital utilization and management of Hirschsprung disease: analysis using the kids' inpatient database. Ann Surg. 2013 Feb;257(2):371-5. doi: 10.1097/SLA.0b013e31827ee976. PMID 23263193
- [Derived] Dharmaraj R, Reno J, Fridge J, Perger L, Zhu Y. Inpatient Care Utilization and Epidemiology of Hirschsprung Disease: Analysis of the National Inpatient Sample. J Pediatr Gastroenterol Nutr. 2022 Jul 1;75(1):3-9. doi: 10.1097/MPG.0000000000003449. Epub 2022 May 27. PMID 35622006